CLINICAL TRIAL: NCT01921738
Title: The Effects of Systemic and Locally Azithromycin Adjunct to Scaling and Root Planning on Clinical and Microbiological Periodontal Indices in Moderate to Severe Chronic Periodontitis
Brief Title: The Effect of Azithromycin in the Treatment of Chronic Periodontitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mahsa Maksabi, Dr, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mnts-o77
Record Dates: First submitted 2013-08-08; First posted 2013-08-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Periodontitis
Keywords: Chronic Periodontitis, Azithromycin, SRP
MeSH Terms: conditions — Chronic Periodontitis | interventions — Azithromycin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1% Azithromycin gel (Experimental): Participants received mechanical periodontal therapy, oral hygiene instructions and placement of the in-situ gel (0.2 ml 1% Azithromycin) into the periodontal pockets in single rooted teeth; twice with an interval of 20 minutes.
  Interventions: Drug: 1% Azithromycin gel
- Azithromycin capsule (Experimental): Participants received mechanical periodontal therapy, oral hygiene instructions and antibiotic (Azithromycin 250mg x 6 capsules)
  Interventions: Drug: Azithromycin
- Placebo Gel (Placebo Comparator): Participants received mechanical periodontal therapy, oral hygiene instructions and placebo (antibiotic) in situ gel.
  Interventions: Drug: placebo gel
- placebo capsule (Placebo Comparator): Participants received mechanical periodontal therapy (Scaling and Root Planing), oral hygiene instructions and placebo (antibiotic) capsules (250mg x 6), at mouth (Po), two times a day (bid) for three days.
  Interventions: Drug: placebo capsule

INTERVENTIONS:
Drug: 1% Azithromycin gel — Participants received mechanical periodontal therapy, oral hygiene instructions and placement of the in-situ gel (0.2 ml 1% Azithromycin) into the periodontal pockets in single rooted teeth; twice with an interval of 20 minutes.
  Other Names: Avindo Gel (Azithromycin Gel 1%); serial number: 8904069410010
  Arms: 1% Azithromycin gel
Drug: Azithromycin — Participants received mechanical periodontal therapy, oral hygiene instructions and antibiotic (Azithromycin 250mg x 6 capsules)
  Other Names: Zithromax (Zimexir, Exir, Brojerd, Iran); serial number: 6260153032097
  Arms: Azithromycin capsule
Drug: placebo gel — Participants received mechanical periodontal therapy, oral hygiene instructions and placebo (antibiotic) in situ gel.
  Other Names: carbopol 934P/974P
  Arms: Placebo Gel
Drug: placebo capsule — Participants received mechanical periodontal therapy (Scaling and Root Planing), oral hygiene instructions and placebo (antibiotic) capsules (250mg x 6), at mouth (Po), two times a day (bid) for three days.
  Other Names: sugar capsule
  Arms: placebo capsule

SUMMARY:
The aim of this study is to investigate the effects of Azithromycin (systemic and locally) on the clinical and microbiological parameters of periodontal in patients with chronic periodontitis.

DETAILED DESCRIPTION:
The double-blind, placebo-controlled clinical trial that is carried out in eighty patients who referred to the Department of Periodontology, Isfahan School of Dentistry. Main inclusion criteria were: 1) Patients with moderate to severe chronic periodontitis 2) At least twenty teeth 3) Age over 18 years. Main exclusion criteria were: 1) History of allergy to the macrolide group 2) History of antibiotic therapy within the 4 months ago 3) The lack of patient cooperation. For all patients is initially performed scaling and root planning (SRP). Oral health education is given to all patients. After one month, patients are randomly divided into four equal groups (two test groups and two control groups). Azithromycin(AZM) 250 milligram (mg) capsules, two times a day (bid), for three days will be given to a test group. In the other test group, 1% AZM gel is locally injected into the periodontal pockets in single-root teeth. Placebo capsules with the same dose and frequency will be given to a control group. In the other control group, placebo gel is injected in the same places. Clinical parameters included pocket depth (PD), clinical attachment level (CAL), papillary bleeding index (PBI), and periodontal disease index (PDI), which are recorded at baseline (before SRP), at 1, 2, 3 and 4 months after treatment. Using polymerase chain reaction (PCR), microbiological assessment of the percentage of Porphyromonas gingivalis (P.g) and Actinobacillus actinomycetemcomitans (A.a) are randomly done for 40 patients (10 patients from each group) at baseline and at 3 months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with moderate to severe chronic periodontitis
2. At least twenty teeth
3. Age over 18 years

Exclusion Criteria:

1. With Systemic diseases that affect periodontal conditions such as: diabetes, blood disorders and diseases of immune system
2. History of antibiotic therapy within the 4 months prior to study
3. History of Allergy to the macrolide group of antibiotics
4. Smoking
5. The lack of patient cooperation
6. History of periodontal treatment during the 4 months prior to the trial
7. Pregnancy
8. Lactating females
9. Patients treated with drugs such as: Anti-acid, Warfarin and Cyclisporine 10) Alcohol use.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Periodontal Pocket Depth | at one, two, three and four months after the intervention.
  measurement was done with color coded periodontal probe (Nordent).
Change from baseline in Clinical Attachment Level | at one, two, three and four months after the intervention.
  measurement was done with color coded periodontal probe (Nordent).
Change from baseline in Modified Gingival Index | at one, two, three and four months after the intervention.
  visual scale, according to Lobene classification.
Change from baseline in Papillary Bleeding Index | at one, two, three and four months after the intervention.
  measurement was done with color coded periodontal probe (Nordent), according to (Muhlemann and Saxer) classification.
Change from baseline in Porphyromonas gingivalis count | at three months after the intervention
  measurement was done with Real Time PCR (Primer Design kits).
Change from baseline in Actinobacillus actinomycetemcomitans count | at three months after the intervention
  measurement was done with Real Time PCR (Primer Design kits).

CONTACTS AND LOCATIONS:
Overall Officials: Mahsa Maksabi, D.D.S, Principal Investigator — Department of Periodontology, Isfahan School of Dentistry
Locations (1):
- School of Dentistry, Isfahan University of Medical Sciences, Isfahan, Isfahan, Iran